CLINICAL TRIAL: NCT00542763
Title: Mycophenolate Sodium Treatment in Patients With Primary Sjogren's Syndrome - An Open Label Pilot Trial
Brief Title: Mycophenolate Sodium Treatment in Patients With Primary Sjogren's Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: myf-01-049
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2007-10-11 (Estimated); Status verified 2004-08

CONDITIONS: Primary Sjogren's Syndrome
Keywords: Sjogren's syndrome; Mycophenolate sodium
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mycophenolate sodium — Medical treatment is initiated with one tablet of 360 mg mycophenolate sodium orally per day for eligible patient. The dosage will be increased weekly by 360 mg up to a maximum stable dose of 1440mg daily. In patients not well tolerating the drug the dosage can be reduced to 720 mg per day.
  Other Names: Myfortic

SUMMARY:
Primary Sjogren's syndrome (pSS) is an autoimmune disorder characterized by keratoconjunctivitis sicca and xerostomia. In addition, various extraglandular manifestations may develop. Several immunomodulating agents have been attempted in the treatment of pSS without achieving satisfactory results. Currently, there is no approved systemic treatment for pSS.

Mycophenolic acid (MPA) is a selective inhibitor of inosine-monophosphate-dehydrogenase which leads to inhibition of the de novo pathway of nucleotide synthesis. The antiproliferative effect of MPA mainly affects activated T- and B-lymphocytes because the proliferation of these cells is critically dependent on the de novo purine synthesis compared to other eukaryotic cells. Since these lymphocytes have been suggested to play a pivotal role in the inflammation and immunopathogenesis of pSS, mycophenolate-sodium might be a promising agent in the treatment of pSS.

We perform a single-centre, open-label pilot trial with Mycophenolate sodium in pSS.

DETAILED DESCRIPTION:
Mycophenolic acid containing compounds such as mycophenolate mofetil and enteric coated mycophenolate sodium are immunosuppressive drugs approved for the prevention of transplant rejection. Mycophenolate mofetil (MMF) is an effective treatment in systemic lupus erythematosus and other autoimmune diseases.

MMF has been used as maintenance therapy after treatment with rituximab (anti-CD20 antibody) in a pSS patient. We have reported a case of successful treatment with MMF in pSS with vasculitis.

The recent observations and the immunosuppressive effect of MPA in other autoimmune diseases led us to evaluate the efficacy and safety of MPA treatment in patients with pSS refractory to other immunosuppressive agents.

The observation period will be 6 months. At baseline, after 3, and after 6 months we examine the clinical status including glandular function tests as well as different laboratory parameters associated with pSS. In addition subjective parameters will be determined on the basis of different questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Sjogren' Syndrome based on the American-European Consensus criteria
* Erythrocyte sedimentation rate >25mm/h and hypergammaglobulinemia (>1500 mg/dl)
* Presence of anti-SS-A and /or SS-B antibodies and / or rheumatoid factor
* Requirement of artificial teardrops due to symptomatic sicca syndrome
* Inadequate response or intolerance of prior treatment with hydroxychloroquine and / or azathioprine
* Adequate contraception for females of childbearing potential

Exclusion Criteria:

* Age below 18 or above 75 years
* Secondary Sjogren's syndrome
* History of cancer, severe infections or other uncontrolled diseases
* Treatment with concomitant disease modifying anti-rheumatic drugs within the least 8 weeks before baseline evaluation
* Prednisolone dose of > 5mg/d or changes of prednisolone dose within the least 4 weeks before baseline
* Use of secretagogues (e.g. pilocarpine, cevimeline) or medications that potentially diminish exocrine gland function (e.g. tricyclic antidepressants, anti-cholinergic drugs)
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of mycophenolate sodium for sicca syndrome and changes in laboratory values associated with the disease | Basline, week 12 and week 24

SECONDARY OUTCOMES:
Safety of mycophenolate sodium in patients with primary Sjogren's syndrome: Clinical examination, full blood count, renal function tests, liver function tests | basline, after week 4, 12, and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Markus Gaubitz, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Mavragani CP, Moutsopoulos NM, Moutsopoulos HM. The management of Sjogren's syndrome. Nat Clin Pract Rheumatol. 2006 May;2(5):252-61. doi: 10.1038/ncprheum0165. PMID 16932698
- [Background] Gaubitz M, Schorat A, Schotte H, Kern P, Domschke W. Mycophenolate mofetil for the treatment of systemic lupus erythematosus: an open pilot trial. Lupus. 1999;8(9):731-6. doi: 10.1191/096120399678840927. PMID 10602445
- [Background] Vitali C, Bombardieri S, Jonsson R, Moutsopoulos HM, Alexander EL, Carsons SE, Daniels TE, Fox PC, Fox RI, Kassan SS, Pillemer SR, Talal N, Weisman MH; European Study Group on Classification Criteria for Sjogren's Syndrome. Classification criteria for Sjogren's syndrome: a revised version of the European criteria proposed by the American-European Consensus Group. Ann Rheum Dis. 2002 Jun;61(6):554-8. doi: 10.1136/ard.61.6.554. PMID 12006334
- [Background] Willeke P, Schotte H, Schluter B, Erren M, Becker H, Dyong A, Mickholz E, Domschke W, Gaubitz M. Interleukin 1beta and tumour necrosis factor alpha secreting cells are increased in the peripheral blood of patients with primary Sjogren's syndrome. Ann Rheum Dis. 2003 Apr;62(4):359-62. doi: 10.1136/ard.62.4.359. PMID 12634239